CLINICAL TRIAL: NCT02852473
Title: Impact of Continuous Positive Airway Pressure on Breathing Motion Amplitude
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erik J. Tryggestad, Ph.D., Associate Professor of Medical Physics, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-001685
Record Dates: First submitted 2016-06-03; First posted 2016-08-02 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Continuous Positive Airway Pressure; Radiotherapy; Proton Therapy
MeSH Terms: conditions — Neoplasms | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Positive Airway Pressure (Experimental): Continuous Positive Airway Pressure (CPAP) will be administered using FDA-approved equipment.
  Interventions: Other: Continuous Positive Airway Pressure

INTERVENTIONS:
Other: Continuous Positive Airway Pressure — CPAP requires subjects to wear a plastic pressurized mask/apparatus, which is connected via a filter and hose to a pump capable of supplying variable pressure (typically on the range of 4-20 cm H2O). The investigators plan to use a full-face mask to prevent subjects from reducing pressure by opening their mouths. If this cannot be tolerated or properly fitted, or is not compatible with the CPAP ventilator, subjects would use a nasal mask only and be asked to keep their mouths closed.

SUMMARY:
This study involves a breathing motion assessment in healthy subjects before and after continuous positive airway pressure (CPAP) administration using MRI images.

The hypothesis for this study is that CPAP administration will significantly reduce breathing motion. This may help cancer patients who are undergoing proton radiotherapy, so they possibly will not have to hold their breath during the procedure.

DETAILED DESCRIPTION:
Minimally invasive techniques for tumor motion reduction that involve free-breathing patients have significant relevance in the context of radiation therapy, in particular proton radiotherapy. Tumor motion reduction has favorable implications for reduction of radiation doses to adjacent healthy organs, radiation plan robustness (accuracy/quality) and for treatment efficiency (reduction of treatment times). Using non-ionizing MRI with volunteers, the investigators will determine the extent to which continuous positive airway pressure (CPAP) reduces breathing motion (diaphragmatic excursion). The researchers will also investigate the parameter space associated with breathing motion reduction versus the amount of pressure applied, as well as timing of initiation of CPAP in relation to the imaging time point (to address whether an initial transient breathing state exists).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult female and males
2. Subject meets routine MRI safety criteria

Exclusion Criteria:

1. Age <18
2. Known history of chronic obstructive pulmonary disease (COPD), asthma, or other chronic pulmonary illness
3. Pregnancy
4. Any safety risk identified via MRI safety screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Breathing Motion Characteristics at High CPAP Setting | Data acquisition for this portion of the study will require approximately 30 minutes.
  Breathing motion at baseline and at initial (higher but tolerable) CPAP settings will be characterized using fast multi-slice, multi-phase 2D gradient-echo or spin-echo MRI sequences in the sagittal or coronal imaging planes over a large field of view covering the thoracic and upper-abdominal region. Specifically "4D-MRI" (or time-resolved MRI) will be generated from retrospective sorting of multi-slice 2D MRI. For these analyses, anatomic reference points (e.g., bright vessels) in multiple organ systems will be identified on the images, contoured or segmented; subsequently 3D motion patterns will be extracted for all anatomical references/features. Numerical simulations will be performed to determine hypothetical radiation target volume changes (cm^3) at these anatomic locations assuming spherical tumors with a given set of tumor diameters (cm).

SECONDARY OUTCOMES:
Change in Breathing Motion Characteristics at Lower CPAP Setting | Approximately 45 minutes into visit.
  Time permitting, the CPAP setting will be reduced to approximately half of the nominal/tolerable/high CPAP setting. Using the same MRI sequences and retrospective sorting technique, 4D-MRI will be generated for this lower CPAP setting. Analogous motion characterization analyses (to outcome measure 1) will be carried out for the lower CPAP setting (relative to baseline 4D-MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Erik J Tryggestad, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided